CLINICAL TRIAL: NCT04620642
Title: Lyon Registry of Stroke Treated by Thrombolysis or Thrombectomy
Acronym: RELATE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0924
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; revascularisation therapy; registry
MeSH Terms: conditions — Ischemic Stroke | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry group: Patients over 18 years old, hospitalized in the neurovascular unit of the Pierre Wertheimer Neurological Hospital (Hospices Civils de Lyon), for an ischemic stroke treated by thrombolysis and / or mechanical thrombectomy and not opposed to this research
  Interventions: Biological: Registry

INTERVENTIONS:
Biological: Registry — No specific intervention. Data of the usual care will be collected as the medical history, the demographic data, the biological analyses, imaging report, etc.

SUMMARY:
This observational study as an objective of characterizing the population of patients treated within the neurovascular unit of the Pierre Wertheimer hospital (Hospices Civils de Lyon) in order to determine their phenotype (age, sex, risk factors, etc.) and its evolution over time. It also aims to assess the management of ischemic stroke (IS) in the neurovascular unit of Pierre Wertheimer Hospital. We will assess in particular the pre-hospital and hospital care times, the type of medical care (thrombolysis and / or thrombectomy) as well as the efficiency of this care (effective recanalization, outcome of patient, etc.).

DETAILED DESCRIPTION:
All patient who has had an IS with an indication of thrombolysis and / or thrombectomy, hospitalized in the neurovascular unit of Pierre Wertheimer Hospital (HCL) since January 2013 and until December 2030 will be contacted for this study

ELIGIBILITY:
Inclusion Criteria:

* - Patients over 18 years old,
* Hospitalization in the neurovascular unit of the Pierre Wertheimer Neurological Hospital (Hospices Civils de Lyon),
* Ischemic stroke treated by thrombolysis and / or mechanical thrombectomy.

Exclusion Criteria:

* - Opposition to this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old, hospitalized in the neurovascular unit of the Pierre Wertheimer Neurological Hospital (Hospices Civils de Lyon), for an ischemic stroke treated by thrombolysis and / or mechanical thrombectomy and not opposed to this research.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Phenotype of the population | 3 months
  Characterization the population of patients with stroke treated by thrombolysis and / or thrombectomy in the neurovascular unit of the Pierre Wertheimer Hospital, Hospices Civils de Lyon : age, sex, risk factors, becoming, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pierre Wertheimer, GHE, HCL, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rascle L, Bani Sadr A, Amaz C, Mewton N, Buisson M, Hermier M, Ong E, Fontaine J, Derex L, Berthezene Y, Eker OF, Cho TH, Nighoghossian N, Mechtouff L. Does the Brush-Sign Reflect Collateral Status and DWI-ASPECTS in Large Vessel Occlusion? Front Neurol. 2022 Mar 2;13:828256. doi: 10.3389/fneur.2022.828256. eCollection 2022. PMID 35309551